CLINICAL TRIAL: NCT05955261
Title: A Collaboration Phase 2 Study of Venetoclax in Combination With Conventional Chemotherapy in Pediatric Patients With Acute Myeloid Leukemia
Brief Title: A Study of Venetoclax in Combination With Conventional Chemotherapy in Pediatric Patients With Acute Myeloid Leukemia
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: PI requests voluntary hold
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML23; NCI-2023-04138 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-06-20; First posted 2023-07-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine; Cytarabine; Gemtuzumab; Daunorubicin; methyl cis-3,4-diamino-2,3,4,6-tetradeoxy-alpha-L-lyxo-hexopyranoside Pt(II); fludarabine phosphate; Idarubicin; Mitoxantrone; Etoposide; gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Risk (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Cytabrine, Danunorubicin Hydrochloride, Gemtuzumab Ozogamicin, Etoposide, Mitoxantrone Hydrochloride, Gilteritinib
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Drug: Daunorubicin Hydrochloride; Drug: Idarubicin Hydrochloride; Drug: Mitoxantrone Hydrochloride; Drug: Etoposide; Drug: Gilteritinib
- Intermediate Risk (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Cytabrine, Danunorubicin Hydrochloride, Fludarabine Phosphate, Gemtuzumab Ozogamicin, Etoposide, Idarubin Hydrochloride, Mitoxantrone Hydrochloride, Gilteritinib
  Interventions: Drug: Venetoclax; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Drug: Daunorubicin Hydrochloride; Drug: Fludarabine Phosphate; Drug: Idarubicin Hydrochloride; Drug: Mitoxantrone Hydrochloride; Drug: Etoposide; Drug: Gilteritinib
- High Risk (Experimental): All eligible patients receive intervention according to the Detailed Description section with the following:
  Venetoclax, Azacitidine, Cytabrine, Danunorubicin Hydrochloride, Fludarabine Phosphate, Gemtuzumab Ozogamicin, Etoposide, Idarubin Hydrochloride, Gilteritinib
  Interventions: Drug: Venetoclax; Drug: Azacitidine; Drug: Cytarabine; Drug: Gemtuzumab Ozogamicin; Drug: Daunorubicin Hydrochloride; Drug: Fludarabine Phosphate; Drug: Idarubicin Hydrochloride; Drug: Etoposide; Drug: Gilteritinib

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be given with each course of therapy. Patients with low-risk AML will receive four courses of therapy, intermediate-risk patients will receive five courses of therapy, and high-risk patients will receive two or three courses of therapy followed by hematopoietic stem cell transplantation.
  Other Names: Venclextra; ABT-99
Drug: Azacitidine — Given IV over 30 minutes on days 1-5
  Other Names: Mylosar; Vidaza
  Arms: High Risk
Drug: Cytarabine — Given IV over 30 minutes q12 hours on days 1-8 (16 doses)
  Other Names: Ara-C; Cytosar-U®
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Mylotarg
Drug: Daunorubicin Hydrochloride — IV over 1 hour on days 1, 3, and 5
  Other Names: FI-6339; L-lyxo-Hexopyranoside
Drug: Fludarabine Phosphate — Given IV over 30 minutes on days 1-5
  Other Names: SH T 586
  Arms: High Risk; Intermediate Risk
Drug: Idarubicin Hydrochloride — Given IV over 15 minutes on days 3-5
  Other Names: IMI-30; Zavedos
Drug: Mitoxantrone Hydrochloride — IV over 1 hour on days 2-4
  Other Names: Neotalem; Pralifan; Novantrone
  Arms: Intermediate Risk; Low Risk
Drug: Etoposide — Given IV over 1 hour on days 1-5
  Other Names: VP-16; Vepesid®
Drug: Gilteritinib — PO on days 8-28 (21 doses)
  Other Names: Xospata

SUMMARY:
This is a phase 2 study to test the hypothesis that venetoclax in combination with standard chemotherapy will be tolerable and active in pediatric patients with newly diagnosed acute myeloid leukemia (AML).

Primary Objectives:

* Establish the tolerability adding venetoclax to standard chemotherapy in pediatric patients with AML
* Estimate the proportion of patients who become minimal residual disease (MRD) negative by flow cytometry after one course of venetoclax-based induction therapy

Secondary Objectives:

- Estimate the rates of complete remission (CR), event-free survival (EFS), and overall survival (OS) in pediatric patients who receive venetoclax-based chemotherapy

DETAILED DESCRIPTION:
Treatment will be based on genetic characteristics and response to therapy. Venetoclax will be given with each course of therapy. Low-risk patients will receive four courses of chemotherapy and intermediate-risk patients will receive five courses. High-risk patients who do not have a suitable stem cell donor or who decline HCT will receive five courses of chemotherapy. The definition of suitable stem cell donor and the conditioning regimens used for HCT will be determined by local institutional protocols or guidelines.

Intervention:

Low Risk

Induction 1: Venetoclax orally (PO) once daily (QD) on days -2 to 11, cytarabine intravenously (IV) over 30 minutes every 12 hours on days 1-8, daunorubicin hydrochloride IV over 1 hour QD on days 1, 3, and 5, etoposide IV over one hour QD on days 1-5, and gemtuzumab ozogamicin IV over 2 hours on day 6.

Induction 2: Venetoclax PO QD on days 1-14, cytarabine IV over 30 minutes every 12 hours on days 1-8, daunorubicin hydrochloride IV over 1 hour QD on days 1, 3, and 5, and etoposide IV over 1 hour QD on days 1-5.

Intensification: Venetoclax PO QD on days 1-7, cytarabine IV over 1-2 hours every 12 hours on days 1-4, and mitoxantrone hydrochloride IV over 1 hour QD on days 2-4 during intensification 1 and then venetoclax PO QD on days 1-7 and high-dose cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5 during intensification 2. Patients with FLT3 activation receive gilteritinib PO QD on days 8-28 during intensification 1 and 2.

Intermediate Risk

Induction 1: Venetoclax orally (PO) once daily (QD) on days -2 to 11, cytarabine intravenously (IV) over 30 minutes every 12 hours on days 1-8, daunorubicin hydrochloride IV over 1 hour QD on days 1, 3, and 5, etoposide IV over one hour QD on days 1-5, and gemtuzumab ozogamicin IV over 2 hours on day 6.

Induction 2: Venetoclax PO QD on days 1-14, fludarabine phosphate IV over 30 minutes QD on days 1-5, cytarabine IV over 3 hours QD starting 4 hours after each dose of fludarabine on days 1-5, idarubicin hydrochloride IV over 15 minutes QD on days 3-5. Patients with FLT3 activation receive gilteritinib PO QD on days 8-28.

Intensification: Venetoclax PO QD on days 1-7, cytarabine IV over 1-2 hours every 12 hours on days 1-4, and mitoxantrone hydrochloride IV over 1 hour QD on days 2-4 during intensification 1, venetoclax PO QD on days 1-7 and high-dose cytarabine IV over 3 hours every 12 hours on days 1, 3, and 5 during intensification 2, and then venetoclax PO QD on days 1-7, cytarabine IV over 1-2 hours every 12 hours on days 1-5, and etoposide IV over 1 hour QD on days 1-5 during intensification 3. Patients with FLT3 activation receive gilteritinib PO QD on days 8-28 during intensification 1-3.

High Risk

Induction 1: Venetoclax orally (PO) once daily (QD) on days -2 to 11, cytarabine intravenously (IV) over 30 minutes every 12 hours on days 1-8, daunorubicin hydrochloride IV over 1 hour QD on days 1, 3, and 5, etoposide IV over one hour QD on days 1-5, and gemtuzumab ozogamicin IV over 2 hours on day 6.

Induction 2: Venetoclax PO QD on days 1-14, fludarabine phosphate IV over 30 minutes QD on days 1-5, cytarabine IV over 3 hours QD starting 4 hours after each dose of fludarabine on days 1-5, idarubicin hydrochloride IV over 15 minutes QD on days 3-5. Patients with FLT3 activation receive gilteritinib PO QD on days 8-28.

Intensification: Patients with MRD < 0.1% proceed directly to HCT if donor is available. If a donor is not yet available, patients with MRD < 0.1% may receive ventoclax PO QD on days 1-21 and azacitidine IV over 30 minutes QD on days 1-5 or venetoclax PO QD on days 1-7, cytarabine IV over 1-2 hours every 12 hours on days 1-5, and etoposide IV over 1 hour QD on days 1-5. Patients with MRD 0.1% to < 1% may receive ventoclax PO QD on days 1-21 and azacitidine IV over 30 minutes QD on days 1-5 or venetoclax PO QD on days 1-7, cytarabine IV over 1-2 hours every 12 hours on days 1-5, and etoposide IV over 1 hour QD on days 1-5. Patients with MRD >= 1% may receive venetoclax PO QD on days 1-10, azacitidine IV over 30 minutes QD on days 1-5, and high-dose cytarabine IV over 3 hours every 12 hours on days 6, 8, and 10. Patients with FLT3 activation receive gilteritinib PO QD on days 8-28.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML fulfilling the criteria of the WHO classification of myeloid neoplasms or < 20% marrow myeloblasts and evidence of a clonal de novo AML genetic abnormality or myeloid sarcoma or primary myelodysplastic syndrome (MDS) with ≥ 10% blasts or a complete blood count with the presence of at least 1,000 blasts/μL (e.g., a WBC count ≥ 10,000/μL with ≥ 10% blasts or a WBC count ≥ 5,000/μL with ≥ 20% blasts
* Age > 28 days and < 22 years
* No prior therapy for this malignancy except for one dose of intrathecal therapy and hydroxyurea or low-dose cytarabine (≤ 200 mg/m^2 per day for ≤ 7 days)
* Female patients of childbearing potential must have a negative pregnancy test within 2 weeks prior to enrollment
* Male and female participants of reproductive potential must agree to use an effective contraceptive method during the study and for 6 months after study treatment
* Written informed consent from the patient and/or parent/legal guardian
* Direct bilirubin ≤ 1.5 x institutional upper limit of normal

Exclusion Criteria:

* Patients with treatment-related AML, Down syndrome, acute promyelocytic leukemia, chronic myeloid leukemia in blast crisis, juvenile myelomonocytic leukemia, Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or other bone marrow failure syndromes are not eligible
* Uncontrolled systemic fungal, bacterial, or viral infection or significant concurrent disease that would compromise patient safety or compliance, study participation, follow up, or interpretation of study results
* Prior exposure to any dose of anthracycline or anthracenedione
* Patients may not receive strong or moderate CYP3A inducers, such as rifampin, within 3 days of enrollment
* Patients may not receive moderate or strong CYP3A inhibitors (e.g., ketoconazole, itraconazole, voriconazole, posaconazole) within 3 days of enrollment.

Ages: 29 Days to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease (MRD)-negativity rate | At day 29 after induction 1
  Will compute a binomial confidence interval for the proportion of MRD-evaluable patients who become MRD-negative (defined as MRD < 0.1%) after induction 1.
Incidence of death or unacceptable adverse event | From initiation to completion of each course of therapy, an average of 6 weeks
  A patient is deemed to have tolerated a course of therapy if they complete that course without death or an unacceptable adverse event. Will monitor the tolerability or each course using multi-stage binomial stopping rules. Will use the method of Jung and Kim to compute 95% confidence intervals that adjust for the multi-stage monitoring.

SECONDARY OUTCOMES:
Event-free survival | From study enrollment to disease resistance, relapse, development of a second malignancy, or death due to any cause (up to 3 years after the last enrollment).
  The Kaplan-Meier method will be used and 95% confidence intervals will be computed for event-free survival at 3 years.
Overall survival | From protocol enrollment until death (up to 3 years after the last enrollment).
  The Kaplan-Meier method will be used and 95% confidence intervals will be computed for overall survival at 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroto Inaba, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (9):
- United States (9):
  - Valley Children's Hospital, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital-San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols